CLINICAL TRIAL: NCT03114514
Title: Efficacy of Platelet-Rich Plasma (PRP) in the Treatment of Periorbital Hyperpigmentation
Brief Title: Efficacy of Platelet-rich Plasma (PRP) in the Treatment of Dark Circles Under the Eyes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UDMS-Dermat-01-2017
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Periorbital Hyperpigmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRP injection (Experimental): A PRP-injection will be performed three times during the course of treatment
  Interventions: Biological: PRP

INTERVENTIONS:
Biological: PRP — PRP will be injected subcutaneously around the eyes at three different time points with one-month interval
  Other Names: platelet-rich plasma

SUMMARY:
10 ml of blood from each patient will be drawn. This blood specimen will be centrifuged in a specific way to get 1 ml of platelet rich plasma (PRP). PRP will be injected into the the skin under the eyes. The treatment course consists of three sessions of PRP injections with one-month intervals between the sessions.

DETAILED DESCRIPTION:
Background:

Dark circles around the eyes is a common problem pretending with relatively dark eyelids concerns many patients, especially women, because of the inconvenience caused by esthetic and negative impact on the psyche and the patient's quality of life. There are several causing factors (such as sun exposure, smoking, alcohol, sleep deprivation, genetic and structural factors). variety of treatments have been used for this situation , but without clear results.

The term 'Platelet-Rich Plasma (PRP)' is a general term used to describe hanging plasma that has been obtained from whole blood with concentration of platelets higher than normal concentration found in the circulating blood. PRP's work mechanism depends on the fact that platelets contain important substances called (growth factors), which have a known role in the process of reform and renewal of tissues.

Aim of the research:

This study was designed to evaluate the effectiveness of (PRP) injection in the treatment of dark circles under the eyes. This is an uncontrolled open therapeutic trial study which will be performed at the Hospital of Dermatology and Venereology of Damascus University in Damascus, Syria during the period from June 2016 to June 2017.

The results will be assessed by standardized digital photography month after each injection and three months after the latest assessment with the assistant of skin colors scale. In addition, the patient's satisfaction with the results and any treatment-related side effects will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with periorbital hyperpigmentation

Exclusion Criteria:

* patients with known platelet dysfunction syndrome
* patients with platelet count less than 100,000 ul
* patient with hemodynamic instability
* patients with severe systemic illness or malignancy or chronic medical illness (e.g. diabetes, chronic infections, and blood dyscrasias).
* patients with local skin disorders or active herpes infection at the site of the procedure.
* patients on anti-coagulants therapy or non-steroidal anti-inflammatory drugs (NSAID) within 48 hours of procedure,
* patients with corticosteroid injection at treatment site within 1 month, systemic use of corticosteroids within 2 weeks
* patients with recent fever or illness, and hemoglobin level< 10 g/dl.
* pregnancy
* history of keloidal scarring.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06-17 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-05-10 (Actual)

PRIMARY OUTCOMES:
Change in Skin Color | Color shade will be measured at one month following the first injection (T1) and at three months following the third injection (T2)
  Standardized digital photographs will be taken and a color scale will be used

SECONDARY OUTCOMES:
Satisfaction | Satisfaction will be measured at three months following the last injection.
  Patients' satisfaction will be measured on a visual analog scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Raed Sameer Noueihed, M.D., Principal Investigator — Resident at the Dermatology and venereology Hospital of Damascus university.
Locations (1):
- Department of Dermatology and Venereology at Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Freitag FM, Cestari TF. What causes dark circles under the eyes? J Cosmet Dermatol. 2007 Sep;6(3):211-5. doi: 10.1111/j.1473-2165.2007.00324.x. PMID 17760701
- [Background] Sheth PB, Shah HA, Dave JN. Periorbital hyperpigmentation: a study of its prevalence, common causative factors and its association with personal habits and other disorders. Indian J Dermatol. 2014 Mar;59(2):151-7. doi: 10.4103/0019-5154.127675. PMID 24700933
- [Background] Roh MR, Chung KY. Infraorbital dark circles: definition, causes, and treatment options. Dermatol Surg. 2009 Aug;35(8):1163-71. doi: 10.1111/j.1524-4725.2009.01213.x. Epub 2009 May 15. PMID 19469797
- [Background] Dohan Ehrenfest DM, Rasmusson L, Albrektsson T. Classification of platelet concentrates: from pure platelet-rich plasma (P-PRP) to leucocyte- and platelet-rich fibrin (L-PRF). Trends Biotechnol. 2009 Mar;27(3):158-67. doi: 10.1016/j.tibtech.2008.11.009. Epub 2009 Jan 31. PMID 19187989
- [Background] Alsousou J, Ali A, Willett K, Harrison P. The role of platelet-rich plasma in tissue regeneration. Platelets. 2013;24(3):173-82. doi: 10.3109/09537104.2012.684730. Epub 2012 May 30. PMID 22647081
- [Background] Sommeling CE, Heyneman A, Hoeksema H, Verbelen J, Stillaert FB, Monstrey S. The use of platelet-rich plasma in plastic surgery: a systematic review. J Plast Reconstr Aesthet Surg. 2013 Mar;66(3):301-11. doi: 10.1016/j.bjps.2012.11.009. Epub 2012 Dec 11. PMID 23238115
- [Background] Abuaf OK, Yildiz H, Baloglu H, Bilgili ME, Simsek HA, Dogan B. Histologic Evidence of New Collagen Formulation Using Platelet Rich Plasma in Skin Rejuvenation: A Prospective Controlled Clinical Study. Ann Dermatol. 2016 Dec;28(6):718-724. doi: 10.5021/ad.2016.28.6.718. Epub 2016 Nov 23. PMID 27904271
- [Background] Conde Montero E, Fernandez Santos ME, Suarez Fernandez R. Platelet-rich plasma: applications in dermatology. Actas Dermosifiliogr. 2015 Mar;106(2):104-11. doi: 10.1016/j.ad.2013.12.021. Epub 2014 May 1. English, Spanish. PMID 24795093